## Colchicine plus Phenolic Monoterpenes to Treat COVID-19 (NCT04392141), 01/20/2021

After collection of data, all continuous variables were presented as the mean ± standard deviation. Categorical variables are presented as N (%). The Kolmogorov–Smirnov test was performed for checking the normality assumption. Moreover, the equality of variance between both groups was tested by Levene's test. After checking the parametric assumptions, Student's t-test (parametric) or the Mann Whitney test (non-parametric) was used to test for statistical differences (two-tailed) between two independent groups. Also paired t-test (parametric) or the Wilcoxon signed-rank test (non-parametric) was used to test for statistical differences between two-time points in each of intervention groups. Two-sided Chi square/Fisher's exact tests were used to assess the associations between intervention groups and the categorical variables. After analyzing the baseline data, using the intention-to-treat (ITT) test, the multiple imputations were conducted by an expectation–maximization (EM) algorithm for making an unbiased comparison between intervention groups in handling missing data. The P-values were not adjusted for multiple testing. All statistical analysis was analyzed using SPSS software (Versions 25). Statistical significance was considered at p<0.05